CLINICAL TRIAL: NCT00318760
Title: Effect of Clonidine on Responses to Imagery Scripts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 999905403; 05-DA-N403
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2014-07-08

CONDITIONS: Cocaine Abuse; Heroin Abuse
Keywords: Drug Cue; Relapse; Stress; Craving
MeSH Terms: conditions — Cocaine-Related Disorders; Heroin Dependence; Recurrence | interventions — Clonidine

ARMS (2):
- ARM 1 (Experimental)
  Interventions: Drug: Clonidine
- ARM 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — 0.1 or 0.2 mg oral, one dose
  Arms: ARM 1
Drug: Placebo — oral capsule 1 dose
  Arms: ARM 2

SUMMARY:
Background:

- Research has shown that clonidine, a drug originally prescribed to treat high blood pressure and some symptoms of opioid withdrawal, can help block stress-induced relapse to heroin and cocaine seeking in rats. However, it does not seem to block cue-induced relapse in rats. Researchers are interested in studying whether clonidine shows the same pattern of effects on stress- and cue-induced cravings for heroin or cocaine in humans.

Objectives:

- To compare the ability of clonidine to reduce stress- and cue-induced cocaine and heroin craving in drug abusers.

Eligibility:

- Individuals between 18 and 55 years of age who are current cocaine or heroin users.

Design:

* This study will consist of two visits: a screening visit to determine eligibility and an experimental/script session.
* Before the script session, participants will provide urine and breath samples for testing. Participants will complete questionnaires to measure their current drug craving and days since last use of cocaine or heroin.
* At the start of the script session, participants will receive a dose of clonidine or placebo as directed by the study researchers. Three hours after dosing, participants will be read four scripts (two neutral, one stress-inducing, and one drug-cue-related) with breaks in between each script. After each script, participants will respond to questions about levels of stress and craving.
* Participants will provide saliva samples immediately before and during the script readings, and will also be measured for skin response to the scripts.

DETAILED DESCRIPTION:
Background. Stress and exposure to drug-related cues (environmental stimuli previously associated with drug availability) are considered factors that increase the risk of relapse to heroin and/or cocaine use. The two factors may act through different neural mechanisms. Alpha-2 adrenergic agonists, such as clonidine, have been shown to block stress-induced relapse, but not cue-induced relapse, to heroin and cocaine self-administration in rodents. The ability of clonidine to attenuate stress- or cue-induced heroin and cocaine craving in drug abusers has not been tested. It is important to determine, in humans, whether clonidine blocks the acute effects of only one putative class of relapse precipitants, or whether its effects are more general.

Scientific goal. To compare the ability of clonidine to reduce stress-induced and cue-induced cocaine and heroin craving in drug abusers.

Participant population. A total of up to 160 drug abusers using cocaine, heroin, or both will be enrolled. Target enrollment will include 40% women and 60% minorities (mostly African-American).

Experimental design and methods. Participants will be randomized to one of three groups receiving clonidine 0.1 mg, clonidine 0.2 mg, or placebo orally under double-blind conditions. The study will consist of a single 5-6 hr experimental session in which there will be baseline measures, drug administration, and four script-guided imagery sets, each followed by a period of data collection. Three hours after dosing (when peak plasma clonidine concentrations are reached), participants will be exposed to four scripts: one stress-inducing, one describing drug cues, and two with neutral content. The standardized script-guided imagery procedure has previously been shown to reliably induce negative affective states (stress scripts) and/or craving (stress and drug-cue scripts) compared to the neutral scripts and to have internal and external validity (Tiffany and Drobes, 1990; Maude-Griffin and Tiffany, 1996; Taylor et al., 2000; Sinha et al., 1999, 2000, 2003; Singleton et al., 2003; Tiffany and Haekeneworth, 1991; Elash et al., 1995; Drobes and Tiffany, 1997; Taylor et al., 2000; Singleton et al., 2003). Outcome measures will include subjective ratings of drug craving and mood, autonomic response (galvanic skin response [GSR]), and endocrine responses (salivary cortisol and salivary ?-amylase, a measure of endogenous adrenergic activity during stress (Chatterton et al., 1996; Nater et al., 2005; van Stegeren et al., 2005)).

Benefits to participants and/or society. There are no direct benefits to participants. However, if clonidine is effective in blocking stress-induced and/or cue-induced craving, then the results will be used as a basis for designing a treatment trial, and drug abusers and society may benefit from the eventual use of clonidine or other alpha agonists for prevention of relapse in cocaine and heroin users. In addition, this research will provide information on the clinical relevance of a preclinical model of relapse, possibly strengthening arguments for its use in medication development.

Risks to participants. Participants may experience side effects from clonidine such as sedation and are expected to experience brief, mild psychological stress and drug craving from the laboratory script procedures. Prior to leaving the session, participants will be assessed for the presence of continued drug effects. If participants are experiencing any stress or craving at the end of the session, they will undergo a 10-minute guided relaxation session, which will be repeated until feelings of stress or craving dissipate, before being released from the laboratory. Participants may be kept longer than the planned session length, up to and including staying overnight on the inpatient ward, because of continued side effects or elevated stress or craving. If the MRP deems it medically necessary, participants will be sent to JHBMC emergency department for further evaluation and treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age between 18 and 55;
  2. Evidence of current cocaine and/or heroin use (by self-report) with a minimum lifetime drug-use duration of 1 year and a minimum current drug use of once in the last 30 days;

     EXCLUSION CRITERIA:

  <!-- -->

  1. Hypersensitivity to clonidine or any component of the formulation
  2. Schizophrenia or any other DSM-IV psychotic disorder; history of anxiety disorder, panic disorder, bipolar disorder; current Major Depressive Disorder
  3. Current physical dependence on opioids, cocaine, alcohol, benzodiazepines or other sedative-hypnotic; this is an exclusion criterion because we want to evaluate the ability of clonidine to affect stress- and cue-induced drug craving independent of its effects on drug withdrawal
  4. Cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires
  5. Pregnancy or breast feeding
  6. Severely impaired hepatic function
  7. Severely impaired renal function, with CLcr < 10 ml/minute
  8. Medical conditions that contraindicate or that could complicate clonidine administration:

     1. hypotension (SBP <95 or DBP < 40 mm Hg) over several readings
     2. hypertension(SBP >160 mm Hg, DBP >95 mm Hg) over several readings
     3. orthostatic hypotension over several readings or as a consequence of any underlying medical disorder (e.g., autonomic insufficiency)
     4. bradycardia (heart rate < 50 bpm) over several readings
     5. cerebrovascular disease or any history of CVA or transient ischemic attack (TIA)
     6. documented coronary disease
     7. serious arrhythmia or conduction defect (e.g., second or third degree heart block, atrial fibrillation)
     8. sinus node dysfunction, severe bradycardia or symptomatic bradycardia
     9. congestive heart failure
  9. Medications that could interact adversely with clonidine: antipsychotics; antihypertensives (e.g., beta blockers); antiepileptics; CNS depressants (e.g. barbiturates, benzodiazepines, narcotic analgesics, alcohol, or other sedatives); cyclosporine; oral hypoglycemic agents or insulin; levodopa; tricyclic antidepressants; herbals such as dong quai, ephedra, yohimbe, ginseng, valerian, St. John s wort, kava kava, gotu kola
  10. Women who are able to get pregnant and are not abstinent from sexual activity must agree to use a medically effective form of contraception while in the study. Those include:

  <!-- -->

  1. Hormonal contraceptives (birth control pills, injectable hormones, vaginal ring hormones),
  2. Surgical sterility (tubal ligation or hysterectomy)
  3. IUD
  4. Diaphragm with spermicide
  5. Condom with spermicide

Women who do not agree to use these medically effective forms of contraception while in the study will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2005-06-14; Study Completion 2013-08-07 (Actual)

PRIMARY OUTCOMES:
Subjective ratings of drug craving and mood | 1 hr
Autonomic response (galvanic skin response [GSR]) | 1 hr
Heart rate and blood pressure | 1 hr
Endocrine responses (salivary cortisol and salivary alpha-amylase) | 1 hr

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie Preston, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Abduljawad KA, Langley RW, Bradshaw CM, Szabadi E. Effects of clonidine and diazepam on the acoustic startle response and on its inhibition by 'prepulses' in man. J Psychopharmacol. 1997;11(1):29-34. doi: 10.1177/026988119701100110. PMID 9097890
- [Background] Benschop RJ, Jacobs R, Sommer B, Schurmeyer TH, Raab JR, Schmidt RE, Schedlowski M. Modulation of the immunologic response to acute stress in humans by beta-blockade or benzodiazepines. FASEB J. 1996 Mar;10(4):517-24. doi: 10.1096/fasebj.10.4.8647351.
- [Background] Berger SP, Hall S, Mickalian JD, Reid MS, Crawford CA, Delucchi K, Carr K, Hall S. Haloperidol antagonism of cue-elicited cocaine craving. Lancet. 1996 Feb 24;347(9000):504-8. doi: 10.1016/s0140-6736(96)91139-3. PMID 8596268